CLINICAL TRIAL: NCT03157817
Title: Sedentary Behaviour, Physical Activity and Cardiometabolic Risk in Chronic Obstructive Pulmonary Disease
Acronym: SPAaRC
Status: Completed | Type: Observational
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Ruth Trethewey, Principal Investigator, Loughborough University
Other Study IDs: SPAaRCLUprotocol1.2
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Obstructive Pulmonary Disease: Patients with a diagnosis of Chronic Obstructive Pulmonary Disease
- Healthy Volunteers: Volunteers without any respiratory condition or symptoms

SUMMARY:
Investigation into the associations between sedentary behaviour, physical activity, body composition and cardiometabolic risk in COPD. A single assessment visit with fasting blood tests, body composition and strength measures followed by a week of activity monitor wear to record sitting time and physical activity. Cardiometabolic risk markers include fasting glucose, HBA1c, HOMA and lipids and blood pressure.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a condition associated with low levels of physical activity and sedentary behaviour (i.e. too much sitting). In addition there is a higher level of heart disease and diabetes in those with COPD. This adds to the burden of the disease. This study will be measuring sitting time using a specific waist-worn monitoring device. The amount of sitting time will then be compared with cardiovascular (heart disease) risk markers, diabetes risk markers and body composition (i.e. fat and muscle mass).

The measurement of cardiovascular and diabetes risk markers will include blood tests to look at blood sugar levels, lipids, cholesterol and insulin resistance as well as blood pressure and heart rate measurement. Body composition measurements will include height, weight, waist circumference, hip circumference as well as scales that will measure body fat and muscle mass and a scan called a dual energy x-ray absorptiometer (DEXA) which uses a type of x-ray to measure body tissues. This involves a very low dose of radiation, much smaller than a normal x-ray.

Quadriceps strength will be measured to provide information on the strength of the muscles.

The sitting device will be worn for 1 week and at the end of this week it will be delivered or sent back by the participant together with a questionnaire about how acceptable the device is to wear.

Additional measures will be included in the assessment in order to examine the results appropriately and reduce bias. These measurements include lung function (breathing) tests, fitness tests (4 metre gait speed and incremental shuttle walk test) and questionnaires about age, gender, ethnicity, medical diagnoses, medications (with detail about oral steroid use), smoking (including pack yrs), exacerbation history, breathlessness, anxiety, depression and motivation, frailty, Physical Activity and Sedentary Behaviour Questionnaire, Employment and Occupational status and history, device Acceptability questionnaire.

Participants will attend an assessment visit. As some of the blood tests need to be done under fasting conditions, i.e. without consuming food or liquids other than water for 8 hours, this will normally take place in the morning. Following the blood tests they will be offered a drink and snack before undertaking any physical measures.

Healthy volunteers of a similar age will also be recruited and attend the same assessment visit to allow comparison between groups to be made.

ELIGIBILITY:
Inclusion Criteria:

1. People with COPD or healthy volunteers without any respiratory conditions
2. Over age of 40
3. Body Mass Index below 35

Exclusion Criteria:

1. Age below 40
2. BMI above 35
3. Unable to complete assessment visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those with COPD recruited from both secondary care and an existing primary care database.
  Healthy volunteers recruited from an existing database recruited through community advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
cardiometabolic risk | baseline
  aggregated measure based on lipid levels, fasting glucose, glycated haemoglobin (A1c) (HbA1c), homeostatic model assessment (HOMA) and blood pressure

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Respiratory Biomedical Research Centre, Leicester, Leicestershire
  - Loughborough Universtiy, Loughborough, Leicestershire

IPD SHARING:
Plan to Share IPD: No
Available on request from Ruth Trethewey